CLINICAL TRIAL: NCT05479097
Title: A Feasibility Study of a Novel mHealth Clinical Decision Support Application to Enable Community Health Workers to Manage Hypertension With Remote Physician Supervision
Brief Title: Feasibility Study of a Novel mHealth Application to Enable Community Health Workers to Manage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Fogarty International Center of the National Institute of Health (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2022-0794; Approval Date 7/2/2022 (Other: UW Madison); A532050 (Other: UW Madison); 1R21TW011891-01 (NIH)
Record Dates: First submitted 2022-07-26; First posted 2022-07-29 (Actual); Results first posted 2024-07-16 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Antihypertensive Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Anti-Hypertensive — Based on information entered by the CHWs into the CommCare application designed for this study, the application will provide recommendations (and underlying rationale for these recommendations) for prescription of antihypertensives (amlodipine and/or losartan OR enalapril) and medications to reduce cardiovascular risk (aspirin and atorvastatin) if indicated, lifestyle modification, and referral to the supervising physician if indicated for potential complications of hypertension.

SUMMARY:
This is a single group study assessing the feasibility of hypertension management by community health workers (CHWs) equipped with a mobile clinical decision support (CDS) application and working with remote physician supervision.

DETAILED DESCRIPTION:
An estimated 1.13 billion people worldwide are currently living with hypertension, the leading preventable cause of death and disability. Two thirds of these patients live in low- and middle-income countries (LMIC). Treatment of hypertension has been found to be cost-effective in reducing morbidity and mortality across a broad range of settings. Despite this, less than 10% of patients with hypertension in LMIC have good control of their blood pressure. Health systems in LMIC, which are often focused on providing episodic care for acute illnesses and suffer from inadequate and poorly distributed health care infrastructure and workforce, are ill-equipped to address the rise in chronic non-communicable diseases (NCDs) such as hypertension. Governments and NGOs are increasingly turning to community health workers (CHWs) - lay people trained to carry out a variety of tasks and who often are from or have a close connection to the communities they serve - to help fill care gaps for hypertension and other NCDs in LMIC. In most cases, CHWs have played supportive (e.g. providing patient education) rather than direct care roles. While such programs have led to improved chronic disease outcomes, they still rely on clinic-based physicians, mid-level providers or nurses to directly provide medical management, and therefore do not address the essential problem of inadequate primary care infrastructure and workforce, particularly in rural areas. Overcoming this problem is key to reducing the growing burden of untreated hypertension in LMIC.

To solve this problem, the investigators are developing an innovative mobile application to assist CHWs in the treatment of hypertension in adults with remote physician supervision. This application is built on the widely-used CommCare platform and will provide clinical decision support (CDS) to CHWs based on protocols from the WHO and the International Society of Hypertension for antihypertensive medication initiation and titration, lifestyle counseling, and identification of patients requiring a higher level of care. The investigators will develop and test this approach in a rural area of Guatemala with poor primary care infrastructure and where the team has worked extensively in the past and has an ongoing collaboration with a local NGO, the San Lucas Mission, and affiliated CHWs. Through this collaboration, the investigators have developed and implemented a CHW-led rural diabetes program enabled by a CDS mobile application and have demonstrated that CHWs can safely and effectively manage diabetes using the application. The hypothesis is that the investigators will be able to adapt the model to hypertension management and are evaluating the feasibility of this approach with this pilot study.

ELIGIBILITY:
Inclusion Criteria:

* Greater than 18 years old
* Diagnosed with hypertension
* Blood pressure greater than or equal to 140/90 mm Hg OR
* currently taking antihypertensive medication

Exclusion Criteria:

* Pregnancy
* Severe comorbid condition(s) with life expectancy less than 1 year

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2023-02-06 (Actual); Primary Completion 2023-08-15 (Actual); Study Completion 2023-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sean Duffy, MD, Principal Investigator — University of Wisconsin-Madison Department of Family Medicine and Community Health
Locations (1):
- San Lucas Mission, San Lucas Tolimán, Departamento de Sololá, Guatemala

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mills KT, Bundy JD, Kelly TN, Reed JE, Kearney PM, Reynolds K, Chen J, He J. Global Disparities of Hypertension Prevalence and Control: A Systematic Analysis of Population-Based Studies From 90 Countries. Circulation. 2016 Aug 9;134(6):441-50. doi: 10.1161/CIRCULATIONAHA.115.018912. PMID 27502908
- [Background] Zhang D, Wang G, Joo H. A Systematic Review of Economic Evidence on Community Hypertension Interventions. Am J Prev Med. 2017 Dec;53(6S2):S121-S130. doi: 10.1016/j.amepre.2017.05.008. PMID 29153113
- [Background] Hunter DJ, Reddy KS. Noncommunicable diseases. N Engl J Med. 2013 Oct 3;369(14):1336-43. doi: 10.1056/NEJMra1109345. No abstract available. PMID 24088093
- [Background] Checkley W, Ghannem H, Irazola V, Kimaiyo S, Levitt NS, Miranda JJ, Niessen L, Prabhakaran D, Rabadan-Diehl C, Ramirez-Zea M, Rubinstein A, Sigamani A, Smith R, Tandon N, Wu Y, Xavier D, Yan LL; GRAND South Network, UnitedHealth Group/National Heart, Lung, and Blood Institute Centers of Excellence. Management of NCD in low- and middle-income countries. Glob Heart. 2014 Dec;9(4):431-43. doi: 10.1016/j.gheart.2014.11.003. PMID 25592798
- [Background] Vedanthan R, Bernabe-Ortiz A, Herasme OI, Joshi R, Lopez-Jaramillo P, Thrift AG, Webster J, Webster R, Yeates K, Gyamfi J, Ieremia M, Johnson C, Kamano JH, Lazo-Porras M, Limbani F, Liu P, McCready T, Miranda JJ, Mohan S, Ogedegbe O, Oldenburg B, Ovbiagele B, Owolabi M, Peiris D, Ponce-Lucero V, Praveen D, Pillay A, Schwalm JD, Tobe SW, Trieu K, Yusoff K, Fuster V. Innovative Approaches to Hypertension Control in Low- and Middle-Income Countries. Cardiol Clin. 2017 Feb;35(1):99-115. doi: 10.1016/j.ccl.2016.08.010. PMID 27886793
- [Background] Kim K, Choi JS, Choi E, Nieman CL, Joo JH, Lin FR, Gitlin LN, Han HR. Effects of Community-Based Health Worker Interventions to Improve Chronic Disease Management and Care Among Vulnerable Populations: A Systematic Review. Am J Public Health. 2016 Apr;106(4):e3-e28. doi: 10.2105/AJPH.2015.302987. Epub 2016 Feb 18. PMID 26890177
- [Background] Mishra SR, Neupane D, Preen D, Kallestrup P, Perry HB. Mitigation of non-communicable diseases in developing countries with community health workers. Global Health. 2015 Nov 10;11:43. doi: 10.1186/s12992-015-0129-5. PMID 26555199
- [Background] Khetan AK, Purushothaman R, Chami T, Hejjaji V, Madan Mohan SK, Josephson RA, Webel AR. The Effectiveness of Community Health Workers for CVD Prevention in LMIC. Glob Heart. 2017 Sep;12(3):233-243.e6. doi: 10.1016/j.gheart.2016.07.001. Epub 2016 Dec 16. PMID 27993594
- [Background] Svoronos T, Mjungu P, Dhadialla R, Luk R, Zue C, Jackson J, et al. CommCare: Automated quality improvement to strengthen community-based health. Weston: D-Tree International 2010
- [Background] Unger T, Borghi C, Charchar F, Khan NA, Poulter NR, Prabhakaran D, Ramirez A, Schlaich M, Stergiou GS, Tomaszewski M, Wainford RD, Williams B, Schutte AE. 2020 International Society of Hypertension Global Hypertension Practice Guidelines. Hypertension. 2020 Jun;75(6):1334-1357. doi: 10.1161/HYPERTENSIONAHA.120.15026. Epub 2020 May 6. No abstract available. PMID 32370572
- [Background] Duffy S, Svenson J, Chavez A, Kelly M, Wise P. Empowering Community Health Workers With Mobile Technology to Treat Diabetes. Ann Fam Med. 2019 Mar;17(2):176. doi: 10.1370/afm.2361. No abstract available. PMID 30858263
- [Background] Duffy S, Norton D, Kelly M, Chavez A, Tun R, Ramirez MNG, Chen G, Wise P, Svenson J. Using Community Health Workers and a Smartphone Application to Improve Diabetes Control in Rural Guatemala. Glob Health Sci Pract. 2020 Dec 23;8(4):699-720. doi: 10.9745/GHSP-D-20-00076. Print 2020 Dec 23. PMID 33361237
- [Derived] Duffy S, Chavez A, Arthur IS, Ortiz GL, Bermudez-Canete A, Nunez-Perez P, White E, Aguilar V, Aguirre J, Dang D, Perez Abaj CS, Letona Lopez YE, Tun R, Valley TM. Feasibility study of a novel mHealth clinical decision support application to enable Community Health Workers to manage hypertension in rural Guatemala. medRxiv [Preprint]. 2026 Jan 23:2026.01.21.26344552. doi: 10.64898/2026.01.21.26344552. PMID 41659079
- See also: World Health Organization. Hypertension Fact Sheet 2019 — https://www.who.int/news-room/fact-sheets/detail/hypertension
- See also: Global Action Plan for the Prevention and Control of NCDs 2013-2020 — https://www.who.int/publications/i/item/9789241506236
- See also: World Health Organization (WHO) HEARTS Technical Package — https://www.knowledge-action-portal.com/en/content/hearts-technical-package
- See also: World Health Organization. Guideline for the pharmacological treatment of hypertension in adults. — https://apps.who.int/iris/bitstream/handle/10665/344424/9789240033986-eng.pdf

RESULTS

PARTICIPANT FLOW:
Groups:
- Study Participants: All study participants were enrolled in a single arm.
Period: Overall Study
Arm/Group | Study Participants
Started | 32
Completed | 30
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Study Participants
Number analyzed (Participants) | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.0 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 32
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 32
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Guatemala | 32
Systolic blood pressure [Median (Inter-Quartile Range); unit: mmHg] | 132.0 [124.8 to 143.5]
Diastolic blood pressure [Mean (Standard Deviation); unit: mmHg] | 80.8 (11.0)

OUTCOME MEASURES:

1. Primary Outcome: Change in Systolic Blood Pressure
Description: Difference in systolic blood pressure from baseline to 6 months
Time Frame: baseline, 6 months
Population: All participants who completed the 6 month follow-up visit
Measure: Median (95% Confidence Interval); unit: mmHg
Arm/Group | Study Participants
Number analyzed (Participants) | 30
mmHg | -7.5 [-12.0 to -1.0]
Statistical Analysis 1: Comparison: Study Participants; The null hypothesis was that there was no change in systolic blood pressure; Test type: Superiority; p = 0.03232, Wilcoxon signed rank test — A priori threshold for statistical significance was P <0.05; Systolic blood pressure was not normally distributed in the study sample, so nonparametric analysis was used; Median Difference (Net) = -7.5, 95% CI 2-sided [-12.0 to -1.0]

2. Primary Outcome: Difference in Diastolic Blood Pressure From Baseline to 6 Months
Description: Difference in diastolic blood pressure from baseline to 6 months
Time Frame: baseline, 6 months
Population: Participants who completed the 6 month visit
Measure: Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Study Participants
Number analyzed (Participants) | 30
mmHg | -3.1 [-6.1 to -0.1]
Statistical Analysis 1: Comparison: Study Participants; The null hypothesis was that there was no change in diastolic blood pressure; Test type: Superiority; p = 0.045, t-test, 2 sided — The a priori threshold for statistical significance was P <0.05; As diastolic blood pressure was normally distributed in our sample, we used a paired t-test to evaluate the mean difference in measurements; Mean Difference (Net) = -3.1, 95% CI 2-sided [-6.1 to -0.1]

3. Primary Outcome: Change in the Proportion of Patients With Systolic Blood Pressure Less Than or Equal to 140
Description: Difference in the proportion of patients with systolic blood pressure less than or equal to 140 from baseline to 6 months
Time Frame: baseline, 6 months
Population: Study participants who completed the 6 month visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Study Participants
Number analyzed (Participants) | 30
Participants
  Baseline systolic blood pressure control: Systolic blood pressure controlled (<=140 mmHg) | 21
  Baseline systolic blood pressure control: Systolic blood pressure not controlled (>140 mmHg) | 9
  Six month systolic blood pressure control: Systolic blood pressure controlled (<=140 mmHg) | 23
  Six month systolic blood pressure control: Systolic blood pressure not controlled (>140 mmHg) | 7
Statistical Analysis 1: Comparison: Study Participants; The null hypothesis was no change in the proportion of patients with systolic blood pressure well-controlled (<=140 mmHg) from baseline to 6 months; Test type: Superiority; p = 0.7237, McNemar — The a priori threshold for statistical significance was P <0.05

4. Primary Outcome: Change in the Proportion of Patients With Systolic Blood Pressure Less Than or Equal to Personalized Goal
Description: Difference in the proportion of patients with systolic blood pressure less than or equal to personalized goal from baseline to 6 months
Time Frame: baseline, 6 months
Population: Participants who completed the 6 month visit. Note that this outcome is the same as outcome #3 (change in proportion of patients with systolic blood pressure <=140 mmHg) because no patients had a personalized goal different than <=140 mmHg.
Measure: Count of Participants; unit: Participants
Arm/Group | Study Participants
Number analyzed (Participants) | 30
Participants
  Baseline: Systolic blood pressure less than or equal to personalized goal | 21
  Baseline: Systolic blood pressure greater than personalized goal | 9
  Six months: Systolic blood pressure less than or equal to personalized goal | 23
  Six months: Systolic blood pressure greater than personalized goal | 7
Statistical Analysis 1: Comparison: Study Participants; The null hypothesis was that there was no difference in the proportion of patients with systolic blood pressure less than or equal to their personalized goal from baseline to 6 months; Test type: Superiority; p = 0.7237, McNemar — The a priori threshold for statistical significance was P <0.05

5. Primary Outcome: Proportion of Visits for Which Both the CHW Conducting the Visit and the Physician Reviewing Post-visit Data Agreed With the Antihypertensive Recommendations Provided by the CDS Application
Description: This measure will be calculated as the proportion of visits for which both the CHW conducting the visit and the physician reviewing post-visit data agreed with the antihypertensive recommendations provided by the application.
Time Frame: 6 months
Measure: Count of Units; unit: Patient visits
Units Other Than Participants: Patient visits
Arm/Group | Study Participants
Number analyzed (Participants) | 32
Number analyzed (Patient visits) | 209
Patient visits
  Visits for which both CHW and physician agreed with medication recommendations | 202
  Visits for which either the CHW or physician disagreed with medication recommendations | 7

ADVERSE EVENTS:
Time Frame: Six months.
Description: Vitals were measured and participants were assessed for medication side effects and potential complications of hypertension at monthly visits using a standardized data collection application. Laboratory testing, including serum creatinine, electrolytes, lipid profile, blood glucose, and ALT was conducted for participants at the enrollment visit and at the 6 month visit, as well as in other points for selected subjects per the medical judgement of the supervising physician.
Arm/Group | Study Participants
All-Cause Mortality (participants affected / at risk) | 0/32
Serious Adverse Events (participants affected / at risk) | 0/32
Other Adverse Events (participants affected / at risk) | 16/32
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study Participants (N=32)
Dyspepsia (Gastrointestinal disorders) | 5 (7)
Non-cardiac chest pain (General disorders) | 4 (6)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (2)
Dizziness (Nervous system disorders) | 2 (2)
Hypotension (Vascular disorders) | 2 (2) — Asymptomatic systolic blood pressure <90 mmHg
Alanine aminotransferase increased (Investigations) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Creatinine increased (Investigations) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1)
Heart failure (Cardiac disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2023-10-02): https://cdn.clinicaltrials.gov/large-docs/97/NCT05479097/Prot_000.pdf
  • Statistical Analysis Plan (2022-04-12): https://cdn.clinicaltrials.gov/large-docs/97/NCT05479097/SAP_001.pdf
  • Informed Consent Form (2023-01-27): https://cdn.clinicaltrials.gov/large-docs/97/NCT05479097/ICF_002.pdf